CLINICAL TRIAL: NCT03313050
Title: A PHASE 1/2, RANDOMIZED, OBSERVER-BLINDED TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A MULTIVALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY ADULTS 50 THROUGH 85 YEARS OF AGE
Brief Title: A Trial To Evaluate A Multivalent Pneumococcal Conjugate Vaccine In Healthy Adults 50-85 Years Of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C3571001
Record Dates: First submitted 2017-10-10; First posted 2017-10-18 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — Vaccines, Combined; Polysaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Observer-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Stage 1 multivalent (ages 50-64 years) (Experimental): multivalent
  Interventions: Biological: Multivalent
- Stage 1 Tdap (ages 50-64 years) (Active Comparator): Tdap
  Interventions: Biological: Tdap
- Stage 2 multivalent (ages 65-85 years) (Experimental): multivalent
  Interventions: Biological: Multivalent
- Stage 2 polysaccharide (ages 65-85 years) (Active Comparator): polysaccharide
  Interventions: Biological: polysaccharide

INTERVENTIONS:
Biological: Multivalent — Pneumococcal conjugate vaccine
  Arms: Stage 1 multivalent (ages 50-64 years); Stage 2 multivalent (ages 65-85 years)
Biological: Tdap — Tetanus, diphtheria, acellular pertussis vaccine
  Arms: Stage 1 Tdap (ages 50-64 years)
Biological: polysaccharide — 23-valent pneumococcal polysaccharide vaccine
  Arms: Stage 2 polysaccharide (ages 65-85 years)

SUMMARY:
This is a 2-stage, phase 1/2, randomized, active-controlled, observer-blinded study with a 2-arm parallel design in each stage.

In Stage 1 healthy adults 50 to 64 years of age with no history of pneumococcal vaccination will be randomized equally to receive either a single intramuscular dose of multivalent pneumococcal conjugate vaccine or a licensed tetanus, diphtheria, acellular pertussis combination vaccine (Tdap) (control group).

In Stage 2 healthy adults 65 to 85 years of age previously vaccinated with Prevnar 13 >=2 months prior to investigational product administration will be randomized equally to receive either a single intramuscular dose of multivalent pneumococcal conjugate vaccine or the licensed 23-valent pneumococcal polysaccharide vaccine (control group).

ELIGIBILITY:
Inclusion Criteria:

* Stage 1: Healthy male or female adults 50 to 64 years of age with no history of pneumococcal vaccination
* Stage 2: Healthy male or female adults 65 to 85 years of age previously vaccinated with Prevnar 13 >= 2 months prior to investigational product administration

Exclusion Criteria:

* Stage 1: Vaccination within 12 months before investigational product administration with diphtheria-, pertussis-, or tetanus-containing vaccine
* Stage 2: Previous vaccination with any pneumococcal vaccine other than a single prior dose of Prevnar 13

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - Achieve Clinical Research LLC, Birmingham, Alabama
  - Core Healthcare Group, Cerritos, California
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Augusta Family Practice, Augusta, Kansas
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Axtell Clinic, P.A., Newton, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Meridian Clinical Research LLC, Omaha, Nebraska
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Omega Medical Research, Warwick, Rhode Island
  - Medical Research South, LLC, Goose Creek, South Carolina
  - J. Lewis Research Incorporated, Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Incorporated/Foothill Family Clinic South, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Essink B, Peterson J, Yacisin K, Lal H, Mirza S, Xu X, Scully IL, Scott DA, Gruber WC, Jansen KU, Watson W. A randomized phase 1/2 study of the safety and immunogenicity of a multivalent pneumococcal conjugate vaccine in healthy adults 50 through 85 years of age. Hum Vaccin Immunother. 2021 Aug 3;17(8):2691-2699. doi: 10.1080/21645515.2021.1890511. Epub 2021 Mar 4. PMID 33661716
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3571001

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1: c7vPnC (50 to 64 Years of Age): In Stage 1, healthy participants aged 50 to 64 years were randomized to receive a single 0.5 milliliter (mL) intramuscular injection of complementary 7-valent pneumococcal conjugate vaccine (c7vPnC) on Day 1. Participants were followed up to 6 months after vaccination.
- Stage 1: Tdap (50 to 64 Years of Age): In Stage 1, healthy participants aged 50 to 64 years were randomized to receive a single 0.5 mL intramuscular injection of tetanus, diphtheria, and acellular pertussis vaccine (Tdap) as control vaccine on Day 1. Participants were followed up to 6 months after vaccination.
- Stage 2: c7vPnC (65 to 85 Years of Age): In Stage 2 healthy participants aged 65 to 85 years, previously vaccinated with Prevnar 13, were randomized to receive a single 0.5 mL intramuscular injection of c7vPnC on Day 1 of Stage 2. Participants were followed up to 12 months after vaccination.
- Stage 2: PPSV23 (65 to 85 Years of Age): In Stage 2, healthy participants aged 65 to 85 years, previously vaccinated with Prevnar 13, were randomized to receive a single 0.5 mL intramuscular injection of 23-valent pneumococcal polysaccharide vaccine (PPSV23 ) as control vaccine on Day 1 of Stage 2. Participants were followed up to 12 months after vaccination.
Period: Stage 1: 6 Months
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age) | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Started | 34 | 32 | 0 | 0
Vaccinated | 34 | 32 | 0 | 0
Completed | 34 | 32 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Stage 2: 12 Months
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age) | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Started | 0 (Stage 1 participants did not continue in Stage 2.) | 0 (Stage 1 participants did not continue in Stage 2.) | 221 (After Stage 1 safety was acceptable then Stage 2 followed with newer participants.) | 224 (After Stage 1 safety was acceptable then Stage 2 followed with newer participants.)
Vaccinated | 0 | 0 | 221 | 223
Completed | 0 | 0 | 210 | 204
Not Completed | 0 | 0 | 11 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 5
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 0 | 3
Not completed — Protocol deviation | 0 | 0 | 7 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of c7vPnC or Tdap or PPSV23 in the study and had post-vaccination follow-up and participants who lacked any safety data were excluded from the analysis.
Groups:
- Stage 1: c7vPnC (50 to 64 Years of Age): In Stage 1, healthy participants aged 50 to 64 years were randomized to receive a single 0.5 mL intramuscular injection of c7vPnC on Day 1. Participants were followed up to 6 months after vaccination.
- Total: Total of all reporting groups
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age) | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age) | Total
Number analyzed (Participants) | 34 | 32 | 221 | 223 | 510
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (4.52) | 58.1 (4.46) | 68.9 (4.72) | 68.8 (3.97) | 67.5 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 131 | 135 | 310
  Male | 11 | 11 | 90 | 88 | 200
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 4 | 10 | 16
  Not Hispanic or Latino | 34 | 30 | 216 | 213 | 493
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 6 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 11 | 9 | 21
  White | 34 | 31 | 204 | 210 | 479
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Percentage of Participants With Local Reactions Within 14 Days After Vaccination
Description: Local reactions included pain at injection site, swelling and redness recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild: greater than (>) 2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm and severe: >10.0 cm. Pain at injection site was graded as mild: did not interfere with activity, moderate: interfered with activity and severe: prevented daily activity.
Time Frame: within 14 days after vaccination
Population: The safety population of Stage 1 included all participants who received at least 1 dose of c7vPnC or Tdap and had post-vaccination follow-up in Stage 1 and participants who lacked any safety data were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age)
Number analyzed (Participants) | 34 | 32
percentage of participants
  Redness: Any | 2.9 [0.1 to 15.3] | 12.5 [3.5 to 29.0]
  Redness: Mild | 2.9 [0.1 to 15.3] | 6.3 [0.8 to 20.8]
  Redness: Moderate | 0 [0.0 to 10.3] | 6.3 [0.8 to 20.8]
  Redness: Severe | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]
  Swelling: Any | 8.8 [1.9 to 23.7] | 18.8 [7.2 to 36.4]
  Swelling: Mild | 5.9 [0.7 to 19.7] | 6.3 [0.8 to 20.8]
  Swelling: Moderate | 2.9 [0.1 to 15.3] | 12.5 [3.5 to 29.0]
  Swelling: Severe | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]
  Pain at injection site: Any | 64.7 [46.5 to 80.3] | 71.9 [53.3 to 86.3]
  Pain at injection site: Mild | 50.0 [32.4 to 67.6] | 59.4 [40.6 to 76.3]
  Pain at injection site: Moderate | 14.7 [5.0 to 31.1] | 12.5 [3.5 to 29.0]
  Pain at injection site: Severe | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]

2. Primary Outcome: Stage 2: Percentage of Participants With Local Reactions Within 14 Days After Vaccination
Description: Local reactions included pain at injection site, swelling and redness recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm. Redness and swelling were graded as mild: >2.0 to 5.0 cm, moderate: >5.0 to 10.0 cm and severe: >10.0 cm. Pain at injection site was graded as mild: did not interfere with activity, moderate: interfered with activity and severe: prevented daily activity.
Time Frame: within 14 days after vaccination
Population: The safety population of Stage 2 included all participants who received at least 1 dose of c7vPnC or PPSV23 and had post-vaccination follow-up in Stage 2 and participants who lacked any safety data were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Number analyzed (Participants) | 221 | 223
percentage of participants
  Redness: Any | 8.1 [4.9 to 12.6] | 17.9 [13.1 to 23.6]
  Redness: Mild | 5.9 [3.2 to 9.8] | 8.1 [4.9 to 12.5]
  Redness: Moderate | 2.3 [0.7 to 5.2] | 4.5 [2.2 to 8.1]
  Redness: Severe | 0 [0.0 to 1.7] | 5.4 [2.8 to 9.2]
  Swelling: Any | 6.8 [3.8 to 10.9] | 16.6 [12.0 to 22.1]
  Swelling: Mild | 5.9 [3.2 to 9.8] | 5.4 [2.8 to 9.2]
  Swelling: Moderate | 0.9 [0.1 to 3.2] | 7.6 [4.5 to 11.9]
  Swelling: Severe | 0 [0.0 to 1.7] | 3.6 [1.6 to 6.9]
  Pain at injection site: Any | 48.4 [41.7 to 55.2] | 61.0 [54.2 to 67.4]
  Pain at injection site: Mild | 46.6 [39.9 to 53.4] | 44.8 [38.2 to 51.6]
  Pain at injection site: Moderate | 1.8 [0.5 to 4.6] | 14.3 [10.0 to 19.6]
  Pain at injection site: Severe | 0 [0.0 to 1.7] | 1.8 [0.5 to 4.5]

3. Primary Outcome: Stage 1: Percentage of Participants With Systemic Events Within 14 Days After Vaccination
Description: Systemic events included fever, fatigue, headache, muscle pain and joint pain recorded by participants in an e-diary. Fever was categorized as: >=38.0 degrees Celsius (C), >=38.0 to 38.4 degrees C, >38.4 to 38.9 degrees C, >38.9 to 40.0 degrees C and >40.0 degrees C. Fatigue, headache, muscle pain and joint pain were graded as any, mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity.
Time Frame: within 14 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age)
Number analyzed (Participants) | 34 | 32
percentage of participants
  Fever: >=38.0 degree C | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]
  Fever: >=38.0 to 38.4 degree C | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]
  Fever: >38.4 to 38.9 degree C | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]
  Fever: >38.9 to 40.0 degree C | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]
  Fever: >40.0 degree C | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]
  Fatigue: Any | 29.4 [15.1 to 47.5] | 28.1 [13.7 to 46.7]
  Fatigue: Mild | 29.4 [15.1 to 47.5] | 9.4 [2.0 to 25.0]
  Fatigue: Moderate | 0 [0.0 to 10.3] | 18.8 [7.2 to 36.4]
  Fatigue: Severe | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]
  Headache: Any | 38.2 [22.2 to 56.4] | 34.4 [18.6 to 53.2]
  Headache: Mild | 23.5 [10.7 to 41.2] | 18.8 [7.2 to 36.4]
  Headache: Moderate | 14.7 [5.0 to 31.1] | 15.6 [5.3 to 32.8]
  Headache: Severe | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]
  Muscle pain: Any | 38.2 [22.2 to 56.4] | 56.3 [37.7 to 73.6]
  Muscle pain: Mild | 26.5 [12.9 to 44.4] | 43.8 [26.4 to 62.3]
  Muscle pain: Moderate | 11.8 [3.3 to 27.5] | 12.5 [3.5 to 29.0]
  Muscle pain: Severe | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]
  Joint pain: Any | 11.8 [3.3 to 27.5] | 15.6 [5.3 to 32.8]
  Joint pain: Mild | 11.8 [3.3 to 27.5] | 12.5 [3.5 to 29.0]
  Joint pain: Moderate | 0 [0.0 to 10.3] | 3.1 [0.1 to 16.2]
  Joint pain: Severe | 0 [0.0 to 10.3] | 0 [0.0 to 10.9]

4. Primary Outcome: Stage 2: Percentage of Participants With Systemic Events Within 14 Days After Vaccination
Description: Systemic events included fever, fatigue, headache, muscle pain and joint pain recorded by participants in an e-diary. Fever was categorized as: >=38.0 degrees C, >=38.0 to 38.4 degrees C, >38.4 to 38.9 degrees C, >38.9 to 40.0 degrees C and >40.0 degrees C. Fatigue, headache, muscle pain and joint pain were graded as any, mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity.
Time Frame: within 14 days after vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Number analyzed (Participants) | 221 | 223
percentage of participants
  Fever: >=38.0 degree C | 0.5 [0.0 to 2.5] | 0.9 [0.1 to 3.2]
  Fever: >=38.0 to 38.4 degree C | 0.5 [0.0 to 2.5] | 0 [0.0 to 1.6]
  Fever: >38.4 to 38.9 degree C | 0 [0.0 to 1.7] | 0.4 [0.0 to 2.5]
  Fever: >38.9 to 40.0 degree C | 0 [0.0 to 1.7] | 0.4 [0.0 to 2.5]
  Fever: >40.0 degree C | 0 [0.0 to 1.7] | 0 [0.0 to 1.6]
  Fatigue: Any | 34.4 [28.1 to 41.1] | 33.2 [27.0 to 39.8]
  Fatigue: Mild | 24.9 [19.3 to 31.1] | 17.5 [12.7 to 23.1]
  Fatigue: Moderate | 7.7 [4.5 to 12.0] | 13.9 [9.6 to 19.1]
  Fatigue: Severe | 1.8 [0.5 to 4.6] | 1.8 [0.5 to 4.5]
  Headache: Any | 24.4 [18.9 to 30.6] | 20.2 [15.1 to 26.1]
  Headache: Mild | 20.4 [15.3 to 26.3] | 14.3 [10.0 to 19.6]
  Headache: Moderate | 3.6 [1.6 to 7.0] | 5.4 [2.8 to 9.2]
  Headache: Severe | 0.5 [0.0 to 2.5] | 0.4 [0.0 to 2.5]
  Muscle pain: Any | 38.5 [32.0 to 45.2] | 46.6 [39.9 to 53.4]
  Muscle pain: Mild | 31.7 [25.6 to 38.2] | 29.1 [23.3 to 35.6]
  Muscle pain: Moderate | 6.3 [3.5 to 10.4] | 16.6 [12.0 to 22.1]
  Muscle pain: Severe | 0.5 [0.0 to 2.5] | 0.9 [0.1 to 3.2]
  Joint pain: Any | 14.9 [10.5 to 20.3] | 19.7 [14.7 to 25.6]
  Joint pain: Mild | 9.5 [6.0 to 14.2] | 12.6 [8.5 to 17.6]
  Joint pain: Moderate | 5.4 [2.8 to 9.3] | 7.2 [4.2 to 11.4]
  Joint pain: Severe | 0 [0.0 to 1.7] | 0 [0.0 to 1.6]

5. Primary Outcome: Stage 1: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both AEs and Non-SAEs.
Time Frame: within 1 month after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age)
Number analyzed (Participants) | 34 | 32
percentage of participants | 8.8 [1.9 to 23.7] | 9.4 [2.0 to 25.0]

6. Primary Outcome: Stage 2: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both AEs and Non-SAEs.
Time Frame: within 1 month after vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Number analyzed (Participants) | 221 | 223
percentage of participants | 10.0 [6.3 to 14.7] | 13.5 [9.3 to 18.6]

7. Primary Outcome: Stage 1: Percentage of Participants With Serious Adverse Events (SAEs) Within 6 Months After Vaccination
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: within 6 months after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age)
Number analyzed (Participants) | 34 | 32
percentage of participants | 5.9 [0.7 to 19.7] | 0 [0.0 to 10.9]

8. Primary Outcome: Stage 2: Percentage of Participants With Serious Adverse Events (SAEs) Within 6 Months After Vaccination
Description: as for outcome 7
Time Frame: within 6 months after vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Number analyzed (Participants) | 221 | 223
percentage of participants | 2.3 [0.7 to 5.2] | 2.7 [1.0 to 5.8]

9. Primary Outcome: Stage 1: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) Within 6 Months After Vaccination
Description: An NDCMC was defined as a disease or medical condition, not previously identified, that is expected to be persistent or is otherwise long-lasting in its effects.
Time Frame: within 6 months after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age)
Number analyzed (Participants) | 34 | 32
percentage of participants | 0 [0.0 to 10.3] | 6.3 [0.8 to 20.8]

10. Primary Outcome: Stage 2: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) Within 6 Months After Vaccination
Description: as for outcome 9
Time Frame: within 6 months after vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Number analyzed (Participants) | 221 | 223
percentage of participants | 3.2 [1.3 to 6.4] | 4.5 [2.2 to 8.1]

11. Primary Outcome: Stage 2: Percentage of Participants With Serious Adverse Events (SAEs) Within 12 Months After Vaccination
Description: as for outcome 7
Time Frame: within 12 months after vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Number analyzed (Participants) | 221 | 223
percentage of participants | 4.1 [1.9 to 7.6] | 3.6 [1.6 to 6.9]

12. Primary Outcome: Stage 2: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) Within 12 Months After Vaccination
Description: as for outcome 9
Time Frame: within 12 months after vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Number analyzed (Participants) | 221 | 223
percentage of participants | 6.8 [3.8 to 10.9] | 6.3 [3.5 to 10.3]

13. Secondary Outcome: Stage 1: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After Vaccination
Description: Antibody-mediated serum OPA against the 7 pneumococcal serotypes specific to c7vPnC (serotypes 8, 10A, 11A, 12F, 15B, 22F and 33F) were measured using a pneumococcal OPA assay. Results were expressed as OPA GMTs. Assay results below the lower limit of quantitation (LLOQ) were set to 0.5*LLOQ in the analysis. Evaluable immunogenicity population = EIP.
Time Frame: 1 month after vaccination
Population: EIP Stage 1:eligible participants with no major protocol deviations, received assigned vaccine, blood collected was within 27-49 days post vaccination, had at least 1 valid and determinate assay result for at least 1 serotype for 1 month after vaccination. 'Number Analyzed' = participants evaluable for this outcome measure at specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age)
Number analyzed (Participants) | 33 | 32
Titer (1/dilution)
  Serotype 8 | 1401 [913.4 to 2147.9] | 16 [9.3 to 26.4]
  Serotype 10A: number analyzed (Participants) | 30 | 28
  Serotype 10A | 6622 [3705.5 to 11833.0] | 92 [35.3 to 239.3]
  Serotype 11A: number analyzed (Participants) | 29 | 30
  Serotype 11A | 3154 [1890.7 to 5262.8] | 604 [302.2 to 1206.4]
  Serotype 12F: number analyzed (Participants) | 25 | 30
  Serotype 12F | 9558 [4114.7 to 22202.0] | 90 [39.6 to 202.8]
  Serotype 15B: number analyzed (Participants) | 28 | 30
  Serotype 15B | 3926 [1526.1 to 10100.2] | 30 [17.9 to 49.7]
  Serotype 22F: number analyzed (Participants) | 30 | 32
  Serotype 22F | 5932 [3625.8 to 9705.6] | 167 [74.4 to 374.3]
  Serotype 33F: number analyzed (Participants) | 27 | 30
  Serotype 33F | 8432 [4116.7 to 17271.3] | 433 [204.7 to 915.4]

14. Secondary Outcome: Stage 2: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titer (GMT) 1 Month After Vaccination
Description: Antibody-mediated serum OPA against the 7 common pneumococcal serotypes specific to c7vPnC (serotypes 8, 10A, 11A, 12F, 15B, 22F and 33F) were measured using a pneumococcal OPA assay. Results were expressed as OPA GMTs. Assay results below the LLOQ were set to 0.5*LLOQ in the analysis.
Time Frame: within 1 month after vaccination
Population: EIP Stage 2:eligible participants with no major protocol deviations, received assigned vaccine, blood collected was within 27-49 days post vaccination, had at least 1 valid and determinate assay result for at least 1 serotype for 1 month after vaccination. Here, 'Number Analyzed' = participants evaluable for this outcome measure at specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Arm/Group | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Number analyzed (Participants) | 219 | 217
Titer (1/dilution)
  Serotype 8: number analyzed (Participants) | 215 | 217
  Serotype 8 | 528 [423.2 to 658.6] | 639 [511.9 to 798.3]
  Serotype 10A: number analyzed (Participants) | 209 | 212
  Serotype 10A | 2297 [1842.9 to 2863.4] | 1052 [802.5 to 1378.9]
  Serotype 11A: number analyzed (Participants) | 215 | 209
  Serotype 11A | 2290 [1854.0 to 2828.7] | 2673 [2182.7 to 3274.6]
  Serotype 12F: number analyzed (Participants) | 210 | 210
  Serotype 12F | 3684 [2926.5 to 4638.6] | 2416 [1852.8 to 3151.0]
  Serotype 15B: number analyzed (Participants) | 216 | 208
  Serotype 15B | 1381 [1019.2 to 1872.2] | 586 [426.0 to 807.2]
  Serotype 22F: number analyzed (Participants) | 211 | 206
  Serotype 22F | 4775 [3889.1 to 5862.2] | 2723 [2123.9 to 3491.1]
  Serotype 33F: number analyzed (Participants) | 209 | 209
  Serotype 33F | 4250 [3403.2 to 5307.2] | 4043 [3082.4 to 5304.3]

15. Secondary Outcome: Stage 1: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rises (GMFRs) From Pre-vaccination to 1 Month After Vaccination
Description: GMFR for the 7 pneumococcal serotypes (serotypes 8, 10A, 11A, 12F, 15B, 22F and 33F) from before Vaccination to one month after Vaccination. Assay results below the LLOQ were set to 0.5*LLOQ in the analysis.
Time Frame: before Vaccination to 1 month after Vaccination
Population: EIP Stage 1:eligible participants with no major protocol deviations, received assigned vaccine, blood collected was within 27-49 days post vaccination, had at least 1 valid and determinate assay result for at least 1 serotype for 1 month after vaccination. Here, 'Number Analyzed' = participants evaluable for this outcome measure at specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age)
Number analyzed (Participants) | 33 | 32
fold rise
  Serotype 8: number analyzed (Participants) | 32 | 31
  Serotype 8 | 106.2 [56.7 to 198.9] | 1.1 [1.0 to 1.3]
  Serotype 10A: number analyzed (Participants) | 29 | 27
  Serotype 10A | 64.7 [28.5 to 146.9] | 1.2 [0.8 to 1.7]
  Serotype 11A: number analyzed (Participants) | 28 | 28
  Serotype 11A | 6.5 [3.0 to 14.2] | 1.0 [0.7 to 1.5]
  Serotype 12F: number analyzed (Participants) | 24 | 29
  Serotype 12F | 261.8 [106.1 to 646.2] | 1.2 [1.0 to 1.4]
  Serotype 15B: number analyzed (Participants) | 28 | 30
  Serotype 15B | 100.2 [32.1 to 312.7] | 1.1 [0.9 to 1.3]
  Serotype 22F: number analyzed (Participants) | 30 | 31
  Serotype 22F | 58.6 [25.0 to 137.3] | 1.4 [1.1 to 1.8]
  Serotype 33F: number analyzed (Participants) | 23 | 24
  Serotype 33F | 27.9 [10.4 to 74.6] | 0.9 [0.6 to 1.5]

16. Secondary Outcome: Stage 2: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rises (GMFRs) From Pre-Vaccination to 1 Month After Vaccination
Description: as for outcome 15
Time Frame: before Vaccination to 1 month after Vaccination
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
Number analyzed (Participants) | 219 | 217
fold rise
  Serotype 8: number analyzed (Participants) | 209 | 212
  Serotype 8 | 30.2 [23.0 to 39.6] | 40.5 [30.4 to 53.8]
  Serotype 10A: number analyzed (Participants) | 200 | 201
  Serotype 10A | 30.6 [21.3 to 43.8] | 15.2 [11.0 to 20.9]
  Serotype 11A: number analyzed (Participants) | 198 | 181
  Serotype 11A | 7.5 [5.6 to 10.1] | 7.0 [5.2 to 9.4]
  Serotype 12F: number analyzed (Participants) | 200 | 196
  Serotype 12F | 64.0 [47.3 to 86.8] | 37.6 [27.2 to 52.0]
  Serotype 15B: number analyzed (Participants) | 210 | 201
  Serotype 15B | 31.7 [22.6 to 44.4] | 16.4 [11.6 to 23.0]
  Serotype 22F: number analyzed (Participants) | 196 | 192
  Serotype 22F | 30.0 [21.1 to 42.7] | 18.6 [13.4 to 25.9]
  Serotype 33F: number analyzed (Participants) | 195 | 194
  Serotype 33F | 10.0 [7.0 to 14.2] | 8.7 [6.3 to 11.9]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events: within 14 days after vaccination; Non serious AEs: Stage 1 and 2- baseline up to 1 month after vaccination (approximately up to 35 days); SAEs: Stage 1- baseline up to 6 months after vaccination (approximately up to 196 days), Stage 2- baseline up to 12 months after vaccination (approximately up to 378 days)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety population evaluated.
Arm/Group | Stage 1: c7vPnC (50 to 64 Years of Age) | Stage 1: Tdap (50 to 64 Years of Age) | Stage 2: c7vPnC (65 to 85 Years of Age) | Stage 2: PPSV23 (65 to 85 Years of Age)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/32 | 3/221 | 0/223
Serious Adverse Events (participants affected / at risk) | 2/34 | 0/32 | 9/221 | 8/223
Other Adverse Events (participants affected / at risk) | 27/34 | 28/32 | 161/221 | 171/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: c7vPnC (50 to 64 Years of Age) (N=34) | Stage 1: Tdap (50 to 64 Years of Age) (N=32) | Stage 2: c7vPnC (65 to 85 Years of Age) (N=221) | Stage 2: PPSV23 (65 to 85 Years of Age) (N=223)
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hernia hiatus repair (Surgical and medical procedures) | 0 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1: c7vPnC (50 to 64 Years of Age) (N=34) | Stage 1: Tdap (50 to 64 Years of Age) (N=32) | Stage 2: c7vPnC (65 to 85 Years of Age) (N=221) | Stage 2: PPSV23 (65 to 85 Years of Age) (N=223)
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 3
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 1
Helicobacter gastritis (Infections and infestations) | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 2
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 33 | 44
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 18 | 85 | 104
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 13 | 11 | 54 | 45
Injection site erythema (General disorders) | 1 | 4 | 18 | 40
Injection site swelling (General disorders) | 3 | 6 | 15 | 37
Fatigue (General disorders) | 10 | 9 | 76 | 74
Injection site pain (General disorders) | 22 | 23 | 107 | 136

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/50/NCT03313050/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT03313050/SAP_001.pdf